CLINICAL TRIAL: NCT04635462
Title: The Cognitive and spOrt Virtual EPIC Training Study: INVESTIGATING THE EFFECTS OF HOME-BASED EXERCISE AND COGNITIVE TRAINING
Brief Title: The Cognitive and spOrt Virtual EPIC Training Study
Acronym: COVEPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Bherer (Other)
Responsible Party: Sponsor-Investigator, Louis Bherer, Associate scientific director, Direction of prevention, Montreal Heart Institute, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-2785
Record Dates: First submitted 2020-11-05; First posted 2020-11-19 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Aging
Keywords: Aging; Remote monitoring; Home-based training; Cognitive Training; Physical Exercise; Cognition
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This clinical trial is a single-blinded study. Research personnel performing the outcome assessments at baseline, three, six and twelve months will be blinded to group allocation. Participants will be aware of the type of training they receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidomain intervention (Experimental): The multidomain intervention will combine a remote monitoring of home-based cognitive training with physical exercise training for 6-month.
  Interventions: Other: Physical exercise training; Other: Cognitive training
- Physical exercise intervention (Experimental): The physical exercises intervention will include the remote monitoring of physical exercise training for 6-month.
  Interventions: Other: Physical exercise training

INTERVENTIONS:
Other: Physical exercise training — Participants will be encouraged to complete exercise training programs in the form of video capsules available via Facebook or Youtube, created by kinesiologists of the Montreal Heart Institut EPIC prevention center. The videos last about 15 minutes and include a warm-up of 3 to 5 minutes, followed a 10-minute training and finally a 2-minute cool-down period. The exercises on video do not require any equipment and integrate, depending on the video, aerobic, muscular strengthening, flexibility and/or balance exercises. Several intensities are described according to the participants' level. Participants will be invited to perform exercise sessions at least 5 times a week, and will be monitored weekly by phone by a member of the research team. The exercise sessions can be performed at home using the video training program, as well as in sports centre or outdoors. For each session, participants have to report its duration, intensity, and the nature of the activity via a follow-up agenda.
Other: Cognitive training — Participants will be encouraged to perform sessions of cognitive training 3 times per week (30 minutes/session). Two of these sessions will involve computer or tablet-based attentional control training targeting dual-tasking, updating and working memory, as well as inhibition and switching. Difficulty of cognitive training will be tailored to participants' performances. The remaining session will consist of memory training. Participants will be instructed different mnemotechnic, as well as be taught about memory in aging in general. The memory training will be provided by videos capsules. To track adherence to cognitive training, participants will be asked to complete a journal and mark days and times where they took part in the various cognitive training sessions.
  Arms: Multidomain intervention

SUMMARY:
The proposed COVEPIC trial is designed to document the effects of remote monitoring of physical exercise and home-based cognitive training on cognitive and physical functions in older adults.

DETAILED DESCRIPTION:
Due to the actual pandemic of COVID-19 around the world, social distancing is recommended, which causes a reduction of social interaction and physical activity. Therefore, this health crisis may have collateral effects on cognitive, physical, and psychological health, especially in elderly people who are more likely to be isolated, and for whom social distancing is of paramount importance. Physical exercise practice has been demonstrated to improve cognitive functioning, along with mobility and physical capacity, and to promote psychological well-being. This is the reason why governmental health authorities, as well as the scientific community recommend to stay physically active, especially in this pandemic period. However, in the current context full-time physical training in sport centres cannot be largely promoted. Effective solutions to help older adults in maintaining regular and efficient physical exercise while maintaining social distancing, are thus needed. Consequently, the current project proposes first to investigate the potential of a remote monitoring of physical activity to promote cognitive, physical and psychological health of older adults. Also, considering the added benefits of combining cognitive training to physical exercise to further enhance health and cognition in seniors, this project also addresses the added benefits of a multidomain intervention combining a physical exercise intervention with a home-based cognitive training.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 50 and older
* Have access to internet
* Have access to a tablet (i.e. iPad or Android) or a computer

Exclusion Criteria:

* Non-cardiopulmonary limitation to exercise (e.g., arthritis)
* Severe exercise intolerance
* Respiratory disease (e.g., asthma, COPD, COVID-19)
* Mini Mental Scale Examination (MMSE) telephone version lower than 19/23
* Diagnostic of cardiovascular disease (e.g., chronic systolic and diastolic heart failure, somatic aortic stenosis, atrial fibrillation, malignant arrhythmias, documented atherosclerotic disease).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Change in general cognitive functioning | Baseline and post-intervention at 6 months.
  Validated remote version of Montreal Cognitive Assessment (0-28 score, with a higher score indicating a better cognitive functioning).
Change in executive functions | Baseline and post-intervention at 6 months.
  Validated remote version of neuropsychological tests and iPad tests (Composite Z-score).
Change in processing speed | Baseline and post-intervention at 6 months.
  Validated remote version of neuropsychological tests and iPad tests (Composite Z-score).
Change in episodic memory | Baseline and post-intervention at 6 months.
  Validated remote version of neuropsychological tests and iPad tests (Composite Z-score).

SECONDARY OUTCOMES:
Change in Walking speed | Baseline and post-intervention at 6 months.
  4-meter walking test (m/s).
Change in Functional mobility | Baseline and post-intervention at 6 months.
  Timed up and Go test (s).
Change in Balance performance | Baseline and post-intervention at 6 months.
  Timed one-leg standing test (s).
Change in Lower limb muscles strength | Baseline and post-intervention at 6 months.
  Timed Sit-to-Stand test (s).
Change in Cardiorespiratory fitness | Baseline and post-intervention at 6 months.
  Matthews cardiorespiratory fitness questionnaire (the score is an estimation of individual VO2 max (ml.kg.min) and range from 15-50, with a higher score indicating a higher VO2max).

OTHER OUTCOMES:
Change in Quality-of-life | Baseline and post-intervention at 6 months.
  36-Item Short Form Health Survey (Scale ranges from 0-100, with a higher score indicating a better health status).
Change in Depressive symptomatology | Baseline and post-intervention at 6 months.
  Geriatric Depression Scale questionnaire (Score ranges from 0-30, with a higher score indicating larger depressive symptomatology).
Change in Anxiety | Baseline and post-intervention at 6 months.
  State-Trait Anxiety Inventory questionnaire (Score ranges from 20-80, with a higher score indicating higher anxiety).
Change in Perceived stress | Baseline and post-intervention at 6 months.
  Perceived Stress Scale questionnaire (Score ranges from 0-4, with 0 no stress,1 mild stress, 3 moderate stress and 4 severe).
Change in Repetitive negative thinking | Baseline and post-intervention at 6 months.
  Perseverative thinking questionnaire (Score ranges from 0-60, with a higher score indicating more repetitive negative thinking).
Change in Self-perceived resilience | Baseline and post-intervention at 6 months.
  Connor-Davidson Resilience Scale 10 questionnaire (Score ranges from 0-40, with a higher indicating better the resilience).
Change in Perceived social support | Baseline and post-intervention at 6 months.
  Lubben Social Network Scale questionnaire (Score ranges from 0-30, with a higher score indicating more social engagement).
Change in Social and community activities involvement | Baseline and post-intervention at 6 months.
  Social and community involvement questionnaire (Score ranges from 0-200, with a higher score indicating more social and community involvement).
Change in Self-reported physical activity | Baseline and post-intervention at 6 months.
  Physical Activity Scale for the Elderly questionnaire (Score ranges from 0-400, with a higher score indicating better level of physical activity).
Change in Sleep quality | Baseline and post-intervention at 6 months.
  Pittsburg Sleep Quality Index questionnaire (Score ranges from 0-21, with a higher score indicating worse sleep quality).
Change in Risk of sleep apnea | Baseline and post-intervention at 6 months.
  Berlin Questionnaire (Participants are classified into High Risk or Low Risk based on their responses to the individual items and their overall scores in the symptom categories.High Risk: if there are 2 or more categories where the score is positive. Low Risk: if there is only 1 or no categories where the score is positive).
Dietary patterns | Baseline.
  Short Diet Questionnaire (Score ranges from 15-45 points, with a score between 15-29 categorised as unhealthy, 30-37 as somewhat unhealthy, and 38 or more as a healthy diet).
Intolerance of Uncertainty | Baseline.
  Intolerance of Uncertainty scale questionnaire (Score ranges from 27-135, with a higher score indicating higher intolerance of uncertainty).
Anxiety Sensitivity | Baseline.
  Anxiety Sensitivity Index questionnaire (Score ranges from 0-64, with a higher score indicating a higher sensitivity to anxiety).
Perceived vulnerability to disease | Baseline.
  Perceived vulnerability to disease questionnaire (Score ranges from 15-95, with a higher score indicating a higher perceived vulnerability to disease).
Cognitive Reserve | Baseline.
  Rami and colleagues' cognitive reserve questionnaire (Scale ranges from 0-26, with a higher score indicating a greater cognitive reserve).
Self-reported masculinity and femininity traits | Baseline.
  Short Form Bem Sex-Role Inventory questionnaire (30 items questionnaire with 10 items assessing the femininity traits, 10 items assessing the masculinity traits, and 10 items neutral, not scored. Two scores are calculated for femininity and masculinity, respectively, and range from 10-70, whit a higher score indicating a higher femininity or masculinity trait).

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bherer, PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Preventive medicine and physical activity centre (centre EPIC), Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooks SK, Webster RK, Smith LE, Woodland L, Wessely S, Greenberg N, Rubin GJ. The psychological impact of quarantine and how to reduce it: rapid review of the evidence. Lancet. 2020 Mar 14;395(10227):912-920. doi: 10.1016/S0140-6736(20)30460-8. Epub 2020 Feb 26. PMID 32112714
- [Background] Jimenez-Pavon D, Carbonell-Baeza A, Lavie CJ. Physical exercise as therapy to fight against the mental and physical consequences of COVID-19 quarantine: Special focus in older people. Prog Cardiovasc Dis. 2020 May-Jun;63(3):386-388. doi: 10.1016/j.pcad.2020.03.009. Epub 2020 Mar 24. No abstract available. PMID 32220590
- [Background] Chen P, Mao L, Nassis GP, Harmer P, Ainsworth BE, Li F. Coronavirus disease (COVID-19): The need to maintain regular physical activity while taking precautions. J Sport Health Sci. 2020 Mar;9(2):103-104. doi: 10.1016/j.jshs.2020.02.001. Epub 2020 Feb 4. No abstract available. PMID 32099716
- [Background] Bherer L, Erickson KI, Liu-Ambrose T. A review of the effects of physical activity and exercise on cognitive and brain functions in older adults. J Aging Res. 2013;2013:657508. doi: 10.1155/2013/657508. Epub 2013 Sep 11. PMID 24102028
- [Background] Colcombe S, Kramer AF. Fitness effects on the cognitive function of older adults: a meta-analytic study. Psychol Sci. 2003 Mar;14(2):125-30. doi: 10.1111/1467-9280.t01-1-01430. PMID 12661673
- [Background] Bherer L. Cognitive plasticity in older adults: effects of cognitive training and physical exercise. Ann N Y Acad Sci. 2015 Mar;1337:1-6. doi: 10.1111/nyas.12682. PMID 25773610
- [Background] Dupuy O, Gauthier CJ, Fraser SA, Desjardins-Crepeau L, Desjardins M, Mekary S, Lesage F, Hoge RD, Pouliot P, Bherer L. Higher levels of cardiovascular fitness are associated with better executive function and prefrontal oxygenation in younger and older women. Front Hum Neurosci. 2015 Feb 18;9:66. doi: 10.3389/fnhum.2015.00066. eCollection 2015. PMID 25741267
- [Background] Renaud M, Bherer L, Maquestiaux F. A high level of physical fitness is associated with more efficient response preparation in older adults. J Gerontol B Psychol Sci Soc Sci. 2010 May;65B(3):317-22. doi: 10.1093/geronb/gbq004. Epub 2010 Feb 5. PMID 20139133
- [Background] Predovan D, Fraser SA, Renaud M, Bherer L. The effect of three months of aerobic training on stroop performance in older adults. J Aging Res. 2012;2012:269815. doi: 10.1155/2012/269815. Epub 2012 Dec 11. PMID 23304504
- [Background] Renaud M, Maquestiaux F, Joncas S, Kergoat MJ, Bherer L. The effect of three months of aerobic training on response preparation in older adults. Front Aging Neurosci. 2010 Nov 11;2:148. doi: 10.3389/fnagi.2010.00148. eCollection 2010. PMID 21151355
- [Background] Lampit A, Hallock H, Valenzuela M. Computerized cognitive training in cognitively healthy older adults: a systematic review and meta-analysis of effect modifiers. PLoS Med. 2014 Nov 18;11(11):e1001756. doi: 10.1371/journal.pmed.1001756. eCollection 2014 Nov. PMID 25405755
- [Background] Gross AL, Parisi JM, Spira AP, Kueider AM, Ko JY, Saczynski JS, Samus QM, Rebok GW. Memory training interventions for older adults: a meta-analysis. Aging Ment Health. 2012;16(6):722-34. doi: 10.1080/13607863.2012.667783. PMID 22423647
- [Background] Ball K, Berch DB, Helmers KF, Jobe JB, Leveck MD, Marsiske M, Morris JN, Rebok GW, Smith DM, Tennstedt SL, Unverzagt FW, Willis SL; Advanced Cognitive Training for Independent and Vital Elderly Study Group. Effects of cognitive training interventions with older adults: a randomized controlled trial. JAMA. 2002 Nov 13;288(18):2271-81. doi: 10.1001/jama.288.18.2271. PMID 12425704
- [Background] Bherer L, Kramer AF, Peterson MS, Colcombe S, Erickson K, Becic E. Training effects on dual-task performance: are there age-related differences in plasticity of attentional control? Psychol Aging. 2005 Dec;20(4):695-709. doi: 10.1037/0882-7974.20.4.695. PMID 16420143
- [Background] Lussier M, Gagnon C, Bherer L. An investigation of response and stimulus modality transfer effects after dual-task training in younger and older. Front Hum Neurosci. 2012 May 18;6:129. doi: 10.3389/fnhum.2012.00129. eCollection 2012. PMID 22629239
- [Background] Payne BR, Stine-Morrow EAL. The Effects of Home-Based Cognitive Training on Verbal Working Memory and Language Comprehension in Older Adulthood. Front Aging Neurosci. 2017 Aug 8;9:256. doi: 10.3389/fnagi.2017.00256. eCollection 2017. PMID 28848421
- [Background] Zhu X, Yin S, Lang M, He R, Li J. The more the better? A meta-analysis on effects of combined cognitive and physical intervention on cognition in healthy older adults. Ageing Res Rev. 2016 Nov;31:67-79. doi: 10.1016/j.arr.2016.07.003. Epub 2016 Jul 14. PMID 27423932
- [Background] Roccaforte WH, Burke WJ, Bayer BL, Wengel SP. Validation of a telephone version of the mini-mental state examination. J Am Geriatr Soc. 1992 Jul;40(7):697-702. doi: 10.1111/j.1532-5415.1992.tb01962.x. PMID 1607586
- [Background] Pendlebury ST, Welch SJ, Cuthbertson FC, Mariz J, Mehta Z, Rothwell PM. Telephone assessment of cognition after transient ischemic attack and stroke: modified telephone interview of cognitive status and telephone Montreal Cognitive Assessment versus face-to-face Montreal Cognitive Assessment and neuropsychological battery. Stroke. 2013 Jan;44(1):227-9. doi: 10.1161/STROKEAHA.112.673384. Epub 2012 Nov 8. PMID 23138443
- [Background] Matthews CE, Heil DP, Freedson PS, Pastides H. Classification of cardiorespiratory fitness without exercise testing. Med Sci Sports Exerc. 1999 Mar;31(3):486-93. doi: 10.1097/00005768-199903000-00019. PMID 10188755
- [Background] Belleville S, Hudon C, Bier N, Brodeur C, Gilbert B, Grenier S, Ouellet MC, Viscogliosi C, Gauthier S. MEMO+: Efficacy, Durability and Effect of Cognitive Training and Psychosocial Intervention in Individuals with Mild Cognitive Impairment. J Am Geriatr Soc. 2018 Apr;66(4):655-663. doi: 10.1111/jgs.15192. Epub 2018 Jan 4. PMID 29313875
- [Derived] Dupuy EG, Besnier F, Gagnon C, Vincent T, Vrinceanu T, Blanchette CA, Gervais J, Breton J, Saillant K, Iglesies-Grau J, Belleville S, Juneau M, Vitali P, Nigam A, Gayda M, Bherer L. Effects of home-based exercise alone or combined with cognitive training on cognition in community-dwelling older adults: A randomized clinical trial. Exp Gerontol. 2024 Dec;198:112628. doi: 10.1016/j.exger.2024.112628. Epub 2024 Nov 9. PMID 39505286
- [Derived] Dupuy EG, Besnier F, Gagnon C, Vincent T, Gregoire CA, Blanchette CA, Saillant K, Bouabdallaoui N, Iglesies-Grau J, Payer M, Marin MF, Belleville S, Juneau M, Vitali P, Gayda M, Nigam A, Bherer L. COVEPIC (Cognitive and spOrt Virtual EPIC training) investigating the effects of home-based physical exercise and cognitive training on cognitive and physical functions in community-dwelling older adults: study protocol of a randomized single-blinded clinical trial. Trials. 2021 Jul 29;22(1):505. doi: 10.1186/s13063-021-05476-2. PMID 34325710